CLINICAL TRIAL: NCT05265806
Title: The Effects of Oxytocin on Social Touch: an fNIRS-based Study
Brief Title: The Effects of Oxytocin Treatment on Social Touch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, : Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-79
Record Dates: First submitted 2022-02-20; First posted 2022-03-04 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: Oxytocin; Social touch; fNIRS
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind mixed experimental design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intranasal oxytocin (Experimental): Participants will be randomly assigned to the administration of oxytocin intranasal spray (24 IU).
  Interventions: Drug: Intranasal oxytocin
- Oral oxytocin (Experimental): Participants will be randomly assigned to the administration of oxytocin lingual spray (24 IU).
  Interventions: Drug: Oral oxytocin
- Placebo (Placebo Comparator): Participants will be randomly assigned to the administration of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal oxytocin — Each subject will be assigned to administration of oxytocin intranasal spray (24 IU).
  Other Names: Oxytocin intranasal spray
  Arms: Intranasal oxytocin
Drug: Oral oxytocin — Each subject will be assigned to administration of oxytocin lingual spray (24 IU).
  Other Names: Oxytocin lingual spray
  Arms: Oral oxytocin
Drug: Placebo — An identical amount of intranasal administration of placebo (identical ingredients except the peptide - i.e. glycerine and sodium chloride) will be assigned to each subject.
  Other Names: PLC
  Arms: Placebo

SUMMARY:
The main aim of the study is to investigate the modulatory effects of oxytocin (24IU) administration on the affective processing of touch manipulated differently in gentle caress-like stroke vs. social massage with a moderate pressure.

DETAILED DESCRIPTION:
A randomized double-blind placebo-controlled mixed experimental design with three arms (intranasal oxytocin administration vs. oral oxytocin administration vs. placebo administration, each with 60 subjects) will be employed in the current study. 35 minutes after treatment subjects will be applied two different types of pleasant touch (social massage vs. caress-like stroking) to their calf. After each applied touch stimulation session, the subjects will be asked to rate their subjective experience of the touch including the perceived pleasantness, arousal, intensity and payment. The neural basis of touch processing will be measured via simultaneously acquired fNIRS together with skin conductance responses and the electrocardiogram recording. Blood samples will be taken before and after the treatment as well as after each run session to measure plasma oxytocin levels to explore the associations with primary outcome measure (the behavioral and neural measures of touch processing). Mixed-measure analysis of variance (ANOVA) with treatment as between-subject factor and condition as within-subject factor will be used to investigate oxytocin effects on social touch processing.

To control potential confounding effects across groups, before the experiment all participants will be asked to complete a range of Chinese versions of validated questionnaires on personality, traits, attitude towards interpersonal touch and sensitivity to reward: Autism Spectrum Quotient (ASQ), Beck Depression Inventory II (BDI), State-Trait Anxiety Inventory (STAI), the Cheek and Buss Shyness Scale (CBSS), the Adult Attachment Scale (AAS), the Childhood Trauma Questionnaire (CTQ), social touch questionnaire (STQ), Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ), Sensory Over-Responsivity (SensOR) Scales and the Interpersonal Reactivity Index (C-IRI). And associations between questionnaire scores (especially the ASQ and STQ scores) with primary outcome measure will be explored to investigate modulatory effects of autistic traits. Additionally, to control for potential confounding effects of treatment on mood across the experiment, the Positive and Negative Affect Schedule (PANAS) will be administered immediately before and 30 minutes after the treatment. Participants will also complete the PANAS after each type of touch condition to further measure the modulatory effects of stroking touch and massage on mood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any past or present psychiatric or neurological disorders and without any current psychotherapeutic medication.

Exclusion Criteria:

* Any history of brain injury, psychiatric/physical illness, alcohol/substance abuse, or other major health concern.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Neural index: fNIRS based measures of touch processing | 35-90 minutes after treatment administration
  fNIRS-based indices of neural processing of social touch after the oxytocin and placebo administration in response to each experimental condition.
Behavioral index: ratings of the pleasantness, arousal, intensity and payment for the applied social touch | 50-90 minutes after treatment administration
  Ratings of perceived pleasantness, arousal, intensity and the willing to pay for the applied caress-like touch and massage after the oxytocin and placebo administration.

SECONDARY OUTCOMES:
Plasma oxytocin concentration | Basal concentration before treatment and altered level during 30-90 minutes after treatment administration
  Basal and altered blood oxytocin concentrations for different treatment groups before and 30 minutes after the administration as well as after each touch condition.
Electrophysiological index: skin conductance responses (SCR) | 35-90 minutes after treatment administration
  SCR amplitudes during touch processing to further investigate oxytocin effects on each experimental condition compared with the placebo.
Electrophysiological index: heart rate variability (HRV) | 35-90 minutes after treatment administration
  HRV reflecting the variability in consecutive heartbeats calculated from electrocardiography during touch processing to further investigate oxytocin effects on each experimental condition compared with the placebo.
Questionnaire scores of autistic traits | Before the experiment
  The Autism Spectrum Quotient (ASQ) scores (0~50, higher scores mean higher autistic trait) to investigate modulatory effects of autistic traits.
Gender difference in the neural and behavioral index | 35-90 minutes after treatment administration
  Gender difference in the neural and behavioral response during the touch processing for different treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Li, Dr., Study Chair — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China(UESTC), Chengdu, Sichuan, China

REFERENCES:
- [Derived] Yamagata T, Ogiwara I, Tatsukawa T, Suzuki T, Otsuka Y, Imaeda N, Mazaki E, Inoue I, Tokonami N, Hibi Y, Itohara S, Yamakawa K. Scn1a-GFP transgenic mouse revealed Nav1.1 expression in neocortical pyramidal tract projection neurons. Elife. 2023 May 23;12:e87495. doi: 10.7554/eLife.87495. PMID 37219072
- [Derived] Chen Y, Zou H, Hou X, Lan C, Wang J, Qing Y, Chen W, Yao S, Kendrick KM. Oxytocin administration enhances pleasantness and neural responses to gentle stroking but not moderate pressure social touch by increasing peripheral concentrations. Elife. 2023 May 12;12:e85847. doi: 10.7554/eLife.85847. PMID 37171081